CLINICAL TRIAL: NCT00408304
Title: Prevention of Depression With Omega-3 Fatty Acids in Chronic Carriers of Hepatitis C Treated With Interferon Alpha.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Schiff1
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2006-12

CONDITIONS: Chronic Hepatitis C
Keywords: interferon alpha; depression; omega 3
MeSH Terms: conditions — Hepatitis C, Chronic; Depression | interventions — Fatty Acids, Omega-3

INTERVENTIONS:
Drug: omega-3 fatty acid

SUMMARY:
The purpose of the study is to check whether development of depression as a side effect of interferon alpha treatment in chronic carriers of hepatitis C can be prevented by omega-3 fatty acids.

DETAILED DESCRIPTION:
Omega-3 fatty acids are known as an alternative treatment for different conditions, including mental conditions, such as depression. We assume that combining omega-3 with the treatment by interferon alpha may prevent the development of depression, which is quite a common side effect of the interferon alpha.

ELIGIBILITY:
Inclusion Criteria:

* Chronic carriers of hepatitis C who start a course of interferon alpha treatment, and are treated in the liver clinic of Bnai Zion hospital.

Exclusion Criteria:

* Disagreement to participation in trial.
* Diagnosed and active mental illness.
* Encephalopathic patients.
* Patients with limited ability to understand the questionnaires or the informed consent process.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-12; Study Completion 2007-12

PRIMARY OUTCOMES:
The effect of omega three fatty acids would be estimated through two questionnaires which filled by the patients monthly
with the BDI questionnaire which estimates the level of depression of the patient and
the SF36 questionnaire which provides information about the overall influence of a disease upon a patient's daily life and mental status.

SECONDARY OUTCOMES:
Secondary outcome measures include monthly results of biochemical and hematologic blood tests, including levels of:
albumin
bilirubin
ALT
CRP
hemoglobin
WBC
platelets

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, MD, Principal Investigator — affiliated with Bnai Zion MC
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel